CLINICAL TRIAL: NCT04771767
Title: Assessing a Combined Ketamine and Online Cognitive Behavioural Therapy Intervention for Treatment Resistant Post-Traumatic Stress Disorder
Brief Title: Combined Ketamine and eCBT Intervention for PTSD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Taras Reshetukha, Principle Investigator, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14521759
Record Dates: First submitted 2020-11-19; First posted 2021-02-25 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Ketamine; Cognitive Behavioral Therapy; Online Cognitive Behavioral Therapy; Pharmacologically enhanced psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with PTSD will be assigned either to the experimental treatment or a control. Data will be collected from participants in both groups at the same 4 time-points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine + eCBT (Experimental): Over 12 weeks, participants receive weekly sessions of asynchronous online cognitive-behavioural therapy as well as 6 sub-anesthetic infusions of Ketamine
  Interventions: Drug: Ketamine; Behavioral: Online Trauma-Focused Cognitive Behavioural Therapy
- Control (No Intervention): Participants are in a control condition receiving treatment as usual, during which time they will not receive the experimental treatment and will have no change in their treatment regimen.

INTERVENTIONS:
Drug: Ketamine — Patients will receive 6 sub-anesthetic IV ketamine infusions over 8 weeks, each one lasting 40 minutes.
  Other Names: Ketalar
  Arms: Ketamine + eCBT
Behavioral: Online Trauma-Focused Cognitive Behavioural Therapy — Participants will enrol in a 12-week online CBT program mirroring in-person trauma-focused CBT.
  Other Names: eCBT; TF-CBT
  Arms: Ketamine + eCBT

SUMMARY:
An open label RCT assessing the efficacy of a combined treatment approach for PTSD, using Ketamine infusions and online Cognitive Behavioural Therapy.

DETAILED DESCRIPTION:
OBJECTIVES

(i) To introduce a previously untreated patient population with PTSD to new therapeutic options.

(ii) To provide new insights into the functional role of Glutamate in affective disorders as well as in learning and memory.

(iii) To explore the utility of pharmacologically-enhanced psychotherapy.

OUTLINE

The present study is an open label randomized control trial assessing the efficacy of a combined treatment of sub-anaesthetic IV Ketamine in conjunction with online CBT (eCBT). In the study, 16 participants with refractory PTSD will be assigned either to an experimental group receiving a combination of Ketamine and eCBT over 12 weeks, or they will be assigned to a 12-week control group. Both groups will be assessed for symptoms of PTSD and comorbid disorders before treatment, at 2 midway points (4 and 8 weeks), and at the end of the 12 week experimental period. Symptoms of PTSD and comorbid disorders for participants in the experimental group are expected to improve significantly more than participants in the control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD by a psychiatrist on the team using the Clinician Administered PTSD Scale (CAPS-5) with a score of at least 50 and a medium presentation.
* Patients will have received at least 2 different types of prior treatment, both of which produced less than a 50% reduction in the participant's symptoms.
* Participants with hypertension or cardiovascular disease must be receiving stable treatment to participate.
* Participants must speak and read English, and will have consistent and reliable access to the internet.
* Patients with suicidal ideation will be included.
* Patients with a history of substance abuse will be included (except for opioid use disorder).

Exclusion Criteria:

Hypomanic/manic episodes, bipolar disorder, acute psychosis, opioid use disorder, treatment with Naltrexone, pregnancy, postpartum, breastfeeding, untreated hypertension, cardiovascular disease, ASPD, active homicidal ideation, and general noncompliance with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Scores on the Clinician Administered PTSD Scale for DSM-5 | 0 weeks from start, 4 weeks from start, 8 weeks from start, and 12 weeks from start
  Assessment of PTSD symptoms for diagnosis and severity; score representing the mildest/lack of symptoms: 0; score representing the most severe symptoms: 120.

SECONDARY OUTCOMES:
Change in Scores on the Montgomery Asberg Depression Rating Scale | 0 weeks from start, 4 weeks from start, 8 weeks from start, and 12 weeks from start
  Measure of depression; score representing the mildest/lack of symptoms: 0; score representing the most severe symptoms: 60.
Change in Scores on the Columbia Suicide Severity Rating Scale | 0 weeks from start, 4 weeks from start, 8 weeks from start, and 12 weeks from start
  Measuring thoughts, feelings, and behaviours associated with suicide; score representing the mildest/lack of symptoms: 0; score representing the most severe symptoms: 6.
Change in Scores on the Sheehan Disabilities Scale | 0 weeks from start, 4 weeks from start, 8 weeks from start, and 12 weeks from start
  A brief, patient rated measure of disability and impairment; score representing the mildest/lack of symptoms: 0; score representing the most severe symptoms: 44.
Change in Scores on the Global Assessment of Functioning | 0 weeks from start, 4 weeks from start, 8 weeks from start, and 12 weeks from start
  Assessing the patient's overall capacity to handle life's challenges; score representing the mildest/lack of symptoms: 100; score representing the most severe symptoms: 1.

CONTACTS AND LOCATIONS:
Overall Officials: Taras Reshetukha, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All participant screening and assessment data will be made available once deidentified.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Made available in June 2024. No end date.
Access Criteria: Open access

REFERENCES:
- [Background] Alavi N, Stefanoff M, Hirji A, Khalid-Khan S. Cognitive Behavioural Therapy through PowerPoint: Efficacy in an Adolescent Clinical Population with Depression and Anxiety. Int J Pediatr. 2018 Nov 8;2018:1396216. doi: 10.1155/2018/1396216. eCollection 2018. PMID 30532790
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Girgenti MJ, Ghosal S, LoPresto D, Taylor JR, Duman RS. Ketamine accelerates fear extinction via mTORC1 signaling. Neurobiol Dis. 2017 Apr;100:1-8. doi: 10.1016/j.nbd.2016.12.026. Epub 2016 Dec 30. PMID 28043916
- [Background] Bisson JI, Roberts NP, Andrew M, Cooper R, Lewis C. Psychological therapies for chronic post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2013 Dec 13;2013(12):CD003388. doi: 10.1002/14651858.CD003388.pub4. PMID 24338345
- [Background] Pradhan B, Mitrev L, Moaddell R, Wainer IW. d-Serine is a potential biomarker for clinical response in treatment of post-traumatic stress disorder using (R,S)-ketamine infusion and TIMBER psychotherapy: A pilot study. Biochim Biophys Acta Proteins Proteom. 2018 Jul;1866(7):831-839. doi: 10.1016/j.bbapap.2018.03.006. Epub 2018 Mar 18. PMID 29563072
- [Derived] Philipp-Muller AE, Reshetukha T, Vazquez G, Milev R, Armstrong D, Jagayat J, Alavi N. Combining Ketamine and Internet-Based Cognitive Behavioral Therapy for the Treatment of Posttraumatic Stress Disorder: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jul 20;10(7):e30334. doi: 10.2196/30334. PMID 34092549